CLINICAL TRIAL: NCT04593758
Title: A Phase I/II Open-Label Trial of CPI-613® (Devimistat) Plus Hydroxychloroquine to Evaluate Maximally Tolerated Dose (MTD), Safety and Efficacy in Patients With Relapsed or Refractory Clear Cell Sarcoma of Soft Tissue
Brief Title: To Evaluate Maximally Tolerated Dose (MTD), Safety and Efficacy of CPI-613® (Devimistat) Plus Hydroxychloroquine in Patients With Relapsed or Refractory Clear Cell Sarcoma of Soft Tissue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCS618
Record Dates: First submitted 2020-10-07; First posted 2020-10-20 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Sarcoma, Clear Cell
MeSH Terms: conditions — Sarcoma, Clear Cell | interventions — devimistat; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613 + Hydroxychloroquine (Experimental): dosing regimen was 600mg hydroxychloroquine PO followed 2 hours later by 2,000 mg/m2 of CPI-613 by central IV infusion over 2 hours followed by 600 mg hydroxychloroquine PO 12 hours following the initial dose daily on days 1 through 5 of every 28 days.
  Interventions: Drug: CPI-613 + Hydroxychloroquine

INTERVENTIONS:
Drug: CPI-613 + Hydroxychloroquine — dosing regimen was 600mg hydroxychloroquine PO followed 2 hours later by 2,000 mg/m2 of CPI-613 by central IV infusion over 2 hours followed by 600 mg hydroxychloroquine PO 12 hours following the initial dose daily on days 1 through 5 of every 28 days.
  Starting dose of 80% of the maximum tolerated (MTD) identified in patients ≥ 45 kg for patients < 45 kg

SUMMARY:
The goal of this trial in Phase I is to determine the maximally tolerated dose (MTD) of hydroxychloroquine in combination with devimistat in patients with relapsed or refractory Clear Cell Sarcomas of the Soft Tissue and to describe the full toxicity profile. In Phase II, the goal is to evaluate the response rate [Complete Rate (CR) + Partial Rate (PR)] of the combination of devimistat and hydroxychloroquine in patients with relapse or refractory Clear Cell Sarcoma of the Soft Tissue and to evaluate the PK and PK/PD profiles for efficacy and safety of the combination of devimistat and hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign the consent. For patients <18yo, consent by a parent or guardian and appropriate assent by the patient will be obtained.
2. Patients must be age ≥ 2 years.
3. Karnofsky performance status ( > 60). For children and adolescent patients, Lansky performance status should be performed and converted to Karnofsky performance status utilizing the conversion table in Appendix IV: Performance Status Conversion Chart.
4. Presence of measurable disease per RECIST v1.1.
5. The phase I portion of the study (dose finding portion) will include patients with relapsed or refractory clear cell sarcoma and other fusion positive relapsed or refractory sarcomas as documented by official pathology report from the diagnosing institution or commercial laboratory.

   Patients with Ewing Sarcoma (EWS) can also be enrolled in the phase I portion of the study only. Patients in the phase 1 portion of the study with EWS will have progressed after at least one prior-line of standard therapy and patients with TRK fusion-positive tumors will have received prior therapy with a TRK inhibitor. Patients must have relapsed or refractory clear cell sarcoma for the phase II portion of the study, defined as a recurrence of disease following or having failed to achieve a response to at least one prior therapy. Diagnosis of clear cell sarcoma must be documented by official pathology report from the diagnosing institution or commercial laboratory including presence of a characteristic translocation such as t(12;22)(q13;q12).
6. Fertile men and their partners who are female of reproductive potential, must agree to abstain from sexual intercourse or to use two highly effective forms of contraception from the time of giving informed consent, during the treatment and for 180 days (females and males) following the last dose of devimistat. A highly effective form of contraception is defined as hormonal oral contraceptives, injectables, patches, intrauterine devices, doublebarrier method (e.g., synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), or male partner sterilization.
7. Organ Function Requirements:

Adequate bone marrow function defined as:

1. For patients with solid tumors without known bone marrow involvement:

   • Peripheral absolute neutrophil count (ANC) ≥ 1,000/mm3

   • Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)

   Adequate Renal Function Defined as:

   • Creatinine clearance or radioisotope GFR ≥ 60mL/min/1.73 m2 or

   • A serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Male Female 2 to < 6 years 0.8 0.8 6 to < 10 years 1.0 1.0 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

   ≥ 16 years 1.7 1.4 The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC.

   Adequate Liver function is defined as:

   • Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age

   • SGPT (ALT) ≤2.5 times the ULN
   * SGOT (AST) ≤2.5 times the ULN
   * Serum albumin ≥ 2 g/dL

   Adequate Neurologic function is defined as:

   • Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled.

   Adequate Blood Pressure.

   Exclusion Criteria:
   1. Have received other chemotherapy within 14 days of initiation of study therapy or immunotherapy (antibody based) within 28 days of initiation of study therapy.
   2. For whom potentially curative anticancer therapy is available.
   3. Are pregnant or breast feeding.
   4. Have known hypersensitivity to any of the components of devimistat or hydroxychloroquine.
   5. Have any other medical or psychological condition, deemed by the physician to be likely to interfere with a subject's ability to sign informed consent, cooperate, or participate in the treatment.
   6. Patients who have an uncontrolled infection are not eligible.
   7. Patients with known G6PD deficiency.
   8. Patients with known underlying retinal disease.
   9. Have immediately life-threatening, severe complications of malignancy such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
   10. Are unable to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of study treatment.
   11. Use of high-risk QT-prolonging drugs and patients with a history of torsades de pointes.
   12. Unresolved toxicity from prior therapy that has failed to resolve to CTCAE ≤ grade 1 or baseline toxicity with the exception of alopecia
   13. History of unstable or deteriorating cardiovascular disease within the previous 6 months prior to screening including but not limited to the following: unstable angina or myocardial infarction, CVA/stroke, Congestive heart failure (New York Heart Association [NYHA] Class III or IV, or uncontrolled clinically significant arrhythmias.
   14. Marked baseline prolongation of QT/QTc interval (repeated exhibition of a QTc interval >480 ms for both male and female patients)
   15. Unwilling or unable to avoid the concomitant use of strong CYP3A4 inducers or inhibitors during study treatment.
   16. Patients concomitantly on tamoxifen are excluded due to increased ocular toxicity with hydroxychloroquine

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
MTD (Phase I) | 6 months
  To determine the maximally tolerated dose (MTD) of hydroxychloroquine in combination with devimistat in mg/m2 based on patient body weight in patients with relapsed or refractory fusion-positive sarcomas and relapsed or refractory clear cell sarcoma.
Toxicity (Phase I) | 6 months
  Dose-limiting toxicities assessed in order to be able to establish the maximum tolerable dose for the combination of CPI-613 and Hydroxychloroquine therapy. Using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 for adverse event reporting (Grade 1 (Mild) - 5 (Death) as well as expectedness (unexpected/expected) and attribution (definitely related to study treatment to unrelated to study treatment).
ORR (Overall Response rate): CR +PR (Phase II) | 12 months
  Overall response rate is defined as the proportion of patients who achieve a best overall response complete response or partial response during or following study treatment

SECONDARY OUTCOMES:
DOR (Duration of Response) | 12 months
  It is the interval from date of initial documented response (CR or PR) to the first documented date of disease progression or death.
PFS (Progression Free Survival) | 12 months
  It is defined as the duration from the date of enrollment to the date of progressive disease or death from any cause.
OS (Overall Survival) | 12 months
  Defines as the time from randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Clevland Clinic, Ohio City, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical Centrer, Nashville, Tennessee
  - Seattle Children's Hospital, Seattle, Washington